CLINICAL TRIAL: NCT00701948
Title: Interest of New Dosages of Inflammatory Markers for the Early Diagnosis of Nosocomial Bacterial Infections of the Newborn
Brief Title: New Dosages of Inflammatory Markers for the Early Diagnosis of Nosocomial Bacterial Infections of the Newborn
Acronym: NOSODIAG
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 4108
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2010-04

CONDITIONS: Nosocomial Infection
Keywords: Late onset neonatal sepsis; Nosocomial bacterial infection; Inflammatory markers; multiplex dosage
MeSH Terms: conditions — Cross Infection; Neonatal Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- A-1: Proven nosocomial bacterial infection (NBI)
- A-2: Possible NBI
- B-1: Absence of NBI
- B-2: Probable absence of NBI

SUMMARY:
This study aims to evaluate new dosage of inflammatory markers or new inflammatory markers for the diagnosis of nosocomial bacterial infection. We made the hypothesis that these new dosages or new inflammatory markers could be more useful than dosage of inflammatory markers already used in clinical practice (especially the use of a combination of interleukins (6 or 8) and C-reactive protein for the management of newborns with a clinical suspicion of nosocomial bacterial infection and especially could allow to avoid excessive treatment with antibiotics

ELIGIBILITY:
Inclusion Criteria:

* Newborns > 72 hours of life hospitalized in neonatal intensive or intermediate care unit presenting a clinical suspicion of NBI

Exclusion Criteria:

* Early post-operative period ( surgery of less than 48 hours)
* Multiple malformations
* Newborn already included in the study for a previous septic events
* Newborn treated with antibiotics in the last 24 hours

Ages: 72 Hours to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborn hospitalized in neonatal intensive care unit with a clinical suspicion of nosocomial bacterial infection
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of new dosage of inflammatory markers or new inflammatory markers for the diagnosis of nosocomial bacterial infection. | 48 hours and at 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Kuhn, MD, Study Director — University Hospital, Strasbourg, France
Locations (2):
- France (2):
  - Service de Pédiatrie 2 - Hôpital d'Enfants CHU de Dijon; 10 - bld Maréchal de Lattre de Tassigny, Dijon
  - Service de Pédiatrie 2 - Hôpital de Hautepierre; 1 - Avenue Molière, Strasbourg